CLINICAL TRIAL: NCT03402191
Title: Comparative Clinical Study Evaluating the Effect of L-arginine Versus Sildenafil in Children With Beta Thalassemia Associated With Pulmonary Hypertension
Brief Title: L-arginine Versus Sildenafil in Children With Beta Thalassemia Associated With Pulmonary Hypertension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, PhDTropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prof Elshanshoury
Record Dates: First submitted 2018-01-09; First posted 2018-01-18 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Thalassemia
MeSH Terms: conditions — Thalassemia | interventions — Arginine; Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- L-arginine (Active Comparator): l-arginine for pulmonary hypertension in patients with thalassemia.
  Interventions: Drug: L-arginine
- Sildenafil (Active Comparator): Sildenafil for pulmonary hypertension in patients with thalassemia.
  Interventions: Drug: Sildenafil
- Control (No Intervention): No pulmonary hypertension

INTERVENTIONS:
Drug: L-arginine — l-arginine for thalassemia with pulmonary hypertension
  Arms: L-arginine
Drug: Sildenafil — Sildenafil for thalassemia with pulmonary hypertension
  Other Names: Viagra
  Arms: Sildenafil

SUMMARY:
This study compares L-arginine Versus Sildenafil as treatment for pulmonary hypertension in Children with Beta Thalassemia

DETAILED DESCRIPTION:
This study focuses on different lines of treatment for pulmonary hypertension in children with thalassemia as this study discusses the Effect of L-arginine Versus Sildenafil in Children with Beta Thalassemia Associated with Pulmonary Hypertension

ELIGIBILITY:
Inclusion Criteria:

* Children with thalassemia and pulmonary hypertension.

Exclusion Criteria:

* Rheumatic heart diseases.
* Other comorbid disease

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with improvement of pulmonary hypertension | 6 months
  patients with improvement of pulmonary hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Sahar El-Haggar, Prof, Principal Investigator — Tanta University - Faculty of Pharmacy; Mohamed El-Shanshoury, Prof, Study Director — Tanta University Pediatrics Department; Osama Abd-rab El-Rasol, Prof, Study Chair — Tanta University Pediatrics Department; Tarek Mostafa, Ass Prof, Study Chair — Tanta University-Faculty of pharmacy; Eman El-Khateeb, Msc, Study Chair — Tanta University-Faculty of pharmacy
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided